CLINICAL TRIAL: NCT04290156
Title: The Effect of Joint Transition Visits on Quality of Life in Adolescents With Inflammatory Bowel Diseases: a Protocol for a Prospective, Randomized, Multicentre, Controlled Trial (TRANS-IBD)
Brief Title: The Effect of Joint Transition Visits on Quality of Life in Inflammatory Bowel Diseases (TRANS-IBD)
Acronym: TRANS-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Sarlós Patrícia, Divison of Gastroenterology, First Department of Medicine, Medical School, University of Pécs, Pécs, Hungary, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50457-2/2019/EKU
Record Dates: First submitted 2020-02-16; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis
Keywords: inflammatory bowel disease; transitional care; adolescents; chronic illness; quality of life; randomized controlled trial
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Chronic Disease

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, two-arm, multicentre trial. The target patient population consists of adolescents with inflammatory bowel diseases (IBD), aged between 16.75 and 17 years. The sample size calculation suggests that 160 subjects (80/ each arm) is required. The allocation ratio is 1:1. Eligible participants in the intervention arm attend a total of four joint transition visits with the adult and the pediatric gastroenterologist. In the control arm, adolescents meet only the pediatric gastroenterologist, but there is a balanced consultation between the two gastroenterologists regarding the patient's treatment plan. Patients in both groups receive the same training and education, the only determinative difference between the two arms is the presence of the adult gastroenterologist at the joint transition visits.
Masking Description: Due to the nature of the study, the blinding of the participants and personnel (pediatric and adult gastroenterologists, medical staff) is not possible, however, the blinding of the data managers and statisticians will be secured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint visits (Experimental): Subjects in the intervention arm attend a total of four joint transition visits performed with the participation of both the adult and the pediatric gastroenterologist.
  Interventions: Other: joint visits
- Usual care (No Intervention): Adolescents meet only the pediatric gastroenterologist, but there is a balanced consultation between the two gastroenterologists with respect the patient's treatment plan.

INTERVENTIONS:
Other: joint visits — The intervention is the implementation of joint transition visits with the participation of both the pediatric and the adult gastroenterologist. One-year intervention period was chosen. In total, there are four joint visits every third months for the adolescents aged 17-18. Each joint visit lasts for at least for 20 minutes, although in case of complex medical history, there is no restriction with respect to the length of the visit. Joint transition visits 1, 2 and 3 (V1-3) are led by the pediatric gastroenterologist, and visit 4 (V4) is led by the adult gastroenterologist.
  Arms: Joint visits

SUMMARY:
Inflammatory bowel diseases (IBD) are among the most common chronic illnesses diagnosed in childhood. Moving from the pediatric to the adult health care is a crucial phase, which can greatly affect adolescents' quality of life. According to the latest international guidelines, based in particular on expert opinions, the implementation of joint visits (involving both pediatric and adult gastroenterologists) are highly recommended during the transition period. This trial aims to prove the beneficial effect of the joint visits.

DETAILED DESCRIPTION:
Transition care is a targeted, well-planned activity, which aims to facilitate the transfer of adolescents with chronic illnesses from pediatric to adult health care. Over the past few years, several recommendations have been introduced with respect to the transitional care of adolescents with inflammatory bowel disease (IBD). According to the international recommendations, joint visits (involving both pediatric and adult gastroenterologists) are highly recommended during the transition period. Although joint visits are considered to be the most optimal form of structured transition, so far, no randomized controlled trial providing strong scientific evidence to prove the superiority of joint visits over usual care has been conducted. TRANS-IBD is a prospective, multicenter, randomized, controlled clinical trial designed to demonstrate the benefits of a structured transitional intervention involving joint visits. Patients in the intervention arm attend a total of four joint visits between the ages of 17 and 18. In the control arm, patients only meet the pediatric gastroenterologist but there is balanced consultation between the adult and the pediatric gastroenterologist, regarding the patient's medical history and treatment plan. Patients in both groups receive the same training and education, the only difference between the two arms is the presence of the adult gastroenterologist at the joint visits. The intervention period of the study starts at the age of 17 and lasts until the age of 18, when the participants are transferred to the adult gastroenterologist. The follow-up period starts from transfer and lasts until the end of the first year spent in the adult gastroenterology care.

ELIGIBILITY:
Inclusion Criteria:

* established IBD diagnosis based on the modified "Porto Criteria" at least 6 months prior to enrolment (date of the diagnostic endoscopy)
* any form of IBD (including Crohn's disease or ulcerative colitis) regardless of disease activity and treatment
* patient aged between 16.75 and 17 years at allocation
* at least one visit attendance at the pediatric gastroenterologist in the year prior to enrolment (aiming to minimize non-adherence with the intervention)
* signed written informed consent from the legal guardian and informed assent from the patients

Exclusion Criteria:

* diagnosis of unclassified IBD (IBD-U)
* pregnancy
* medically certified developmental or intellectual disabilities (when it is expected that the patient is unable to fill the questionnaires)
* history of cancer or active cancer treatment
* BMI ≥ 40
* concomitant participation in another interventional clinical trial
* conditions when follow-up cannot be fulfilled (e.g., plan for studying or working abroad after the age of 18)

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported health-related quality of life (HRQoL) one year after transfer | 24 months
  HRQoL is measured with a validated and IBD-specific questionnaire, called IMPACT III (HR) (unabbreviated scale title is not existing). It consists of 35-items, using a five-point Likert self-completed response scale. The questions are related to the severity and frequency of the following symptoms over the last two weeks: bowel symptoms, systemic symptoms, emotional functioning, social functioning, body image and treatments or interventions. The lowest score is 35, that can be achieved, and the maximum is 175 points. Higher scores indicate better HRQoL.

SECONDARY OUTCOMES:
The number of patients not lost to follow-up | 24 months
  Patients are considered as not lost to follow-up if they attend at least three out of the five planned visits with the adult gastroenterologist (AGE) during the follow-up period. Previously cancelled and then rescheduled AGE visits are acceptable.
Medication adherence | 24 months
  Measured with the Medical Adherence Report Scale (MARS-5) which consist of five statements with respect to the patient's medical adherence in the last one week. Patients can describe their behavior on a five-point Likert response scale ranging from 'always' to 'never' (1-5 points). The lowest total score that can be achieved is 5 (lowest adherence), while the highest is 25 (maximal adherence). Higher scores indicate better medical adherence.
Self-efficacy: IBDSES-A | 24 months
  Measured with IBD Self-Efficacy Scale for adolescents and young adults (IBDSES-A) questionnaire, which investigates the person's confidence in their ability to manage demands and is predictive of health outcomes in chronic disease. The maximum scores range from 21 to 57 (as reverse scoring is used in case of 2 items). Higher scores indicate higher self-efficacy.
Patient's satisfaction: CACHE | 24 months
  Measured with CACHE questionnaire (unabbreviated scale title is not existing), which consists of 31 questions with respect to the attitude of the medical team, the location, accessibility, and facilities of the IBD centre. Questions can be answered with a five-point Likert response scale. The final score can be given on a scale that ranges from 0 (minimum satisfaction) to 100 (maximum satisfaction). The final total score is calculated with standardization, using the following formula to determine the points of each individual item: (real score-minimum score)/ (maximum score-minimum score) ×100. Higher score indicates higher level of satisfaction.
Transition readiness (1) | 24 months
  Transition readiness is measured with the validated tool of Transition Readiness Questionnaire (STARx). STARx consists of three modules (with a total of 18 items), aiming to investigate the sense of responsibility, the disease-specific knowledge and the independency of the patients. Each item can be answered using a five-point Likert response scale and can be scored between 1 and 5 points. The maximum score is 90, higher score indicates better transition readiness. STARx is filled out by the participating adolescents and by their legal guardian too.
Transition readiness (2) | 24 months
  Transition readiness is measured with the validated tool of Transition Readiness Assessment Questionnaire (TRAQ). TRAQ consisting of 20 items and assesses the adolescents' willingness to be involved in or to be completely independent in managing disease related tasks (e.g., taking medications, making appointments, getting medications prescribed). A five-point Likert response scale (with scores range from 1 to 5) is used for answering each question. A total of 100 point can be acquired. In case of both tool, higher total scores indicate a higher level of transition readiness.
The number of flare-ups | 24 months
  Flare-ups are defined as clinical symptoms suggesting disease activity, accompanied with biochemical (e.g., stool calprotectin, c-reactive protein (CRP)), endoscopic, or imaging evidence of inflammation. Intensifying disease symptoms resulting in dose escalation or initiation of a new drug aiming to achieve remission are also considered as flare-ups.
The number of patients who needed the initiation of corticosteroid treatment | 24 months
  The number of patients who needed the initiation of corticosteroid treatment including the initiation of topical and systemic steroid formulations
The number of patients who needed the initiation of biological treatment | 24 months
  The number of patients who needed the initiation of biological treatment including the initiation of all types of biologics registered for the treatment of IBD
Stool calprotectin level | 24 months
  Measured in unit: mg/g
Disease activity (1) | 24 months
  In case of Crohn's disease, Pediatric Crohn's Disease Activity Index (PCDAI) is being used for the assessment of disease activity. PCDAI counts with clinical symptoms (e. g. abdominal pain, stool frequency) and laboratory parameters (e.g.: haematocrit, erythrocyte sedimentation rate, serum albumin level).
  The minimum of 0 point can be achieved, while the maximum is 110 points. Higher score indicates higher disease activity. (<10 points: Remission; 11-30 points: Moderate disease activity; >31 points: Severe disease activity)
Disease activity (2) | 24 months
  In case of Ulcerative Colitis, Pediatric Ulcerative Colitis Activity Index (PUCAI) is being used for the assessment of disease activity. PUCAI counts with clinical symptoms (e.g. abdominal pain, rectal bleeding, and activity level).
  The minimum of 0 point can be achieved, while the maximum is 85 points. Higher score indicates higher disease activity. (<10 points: Remission; 11-30 points: Moderate disease activity; >31 points: Severe disease activity)
Disease activity (3) | 24 months
  In case of luminal Crohn's disease, Crohn's Disease Activity Index (CDAI) is being used for the assessment of disease activity. CDAI is the sum of eight components (clinical symptoms (e.g. abdominal pain, number of liquid stools), finding of the physical examination (e.g. abdominal mass, body weight), laboratory parameters (e.g. Haematocrit)) to each of which is assigned a specific weight.
  The minimum of 0 point can be achieved, while the maximum is 600 points. Higher score indicates higher disease activity. (<150 points: Inactive disease; 151-220 points: Mild disease activity; 221-300: Moderate disease activity; 301-450: Severe disease activity; >450: Fulminant disease activity)
Disease activity (4) | 24 months
  In case of perianal Crohn's disease perianal Crohn's Disease Activity Index (pCDAI) is being used for the assessment of disease activity. pCDAI counts with the discharge, the pain/ restrictions of activities, the restrictions of sexual activities, and with the type of perianal disease.
  The minimum of 0 point can be achieved, while the maximum is 20 points. Higher score indicates higher perianal disease activity.
Disease activity (5) | 24 months
  In case of Ulcerative Colitis Mayo score is being used for the assessment of disease activity. Mayo score clinical symptoms (e.g. abdominal pain, rectal bleeding), findings of the endoscopy, and the physician's global assessment).
  The minimum of 0 point can be achieved, while the maximum is 12 points. Higher score indicates higher disease activity. (0-3 points: inactive disease, 4-6 points: mild disease activity, 7-9 points: moderate disease activity, >9 points: severe disease activity)
Laboratory parameter refers to inflammation: C-reactive protein (CRP) | 24 months
  C-reactive protein (CRP) is measured in unit: mg/l. Higher value of CRP indicates greater inflammation.
Laboratory parameter refers to inflammation: White blood cell count (WBC) | 24 months
  White blood cell count (WBC) is measured in unit: G/L. Higher value of WBC indicates greater inflammation.
Laboratory parameter refers to inflammation: Erythrocyte sedimentation rate (ESR) | 24 months
  Erythrocyte sedimentation rate (ESR) is measured in unit: mm/hour. Higher value of ESR indicates greater inflammation.
The number of unplanned visits at the caregiver gastroenterologist | 24 months
  Medical visits, which were not arranged in advance with the caring gastroenterologist, are considered unplanned visits
The number of visits at the emergency department | 24 months
  The number of visits at the emergency department, which are needed due to acute severe symptoms of IBD
The number of scheduled imaging performed | 24 months
  The number of images including abdominal ultrasound, x-ray, MRI, CT-scan and other images, which were arranged in advance
The number of urgent imaging performed | 24 months
  The number of images including abdominal ultrasound, x-ray, MRI, CT-scan and other images, which were not arranged in advance
The number of scheduled endoscopies performed | 24 months
  The number of endoscopies including gastroduodenoscopy and colonoscopy, which were arranged in advance
The number of urgent endoscopies performed | 24 months
  The number of endoscopies including gastroduodenoscopy and colonoscopy, which were not arranged in advance
The number of IBD-related surgical interventions performed | 24 months
  The number of surgical interventions, which were performed because of IBD
The number of IBD related hospital admissions | 24 months
  The number of hospital admissions, which were needed because of IBD
The length of IBD-related hospitalization | 24 months
  The length of the IBD-related hospitalization given in days.

CONTACTS AND LOCATIONS:
Overall Officials: Péter Hegyi, MD, PhD, DSc, Study Chair — Insitute for Translational Medicine, University of Pécs, HU; Patrícia Sarlós, MD, PhD, Principal Investigator — First Department of Medicine, University of Pécs, Medical School, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks AJ, Smith PJ, Cohen R, Collins P, Douds A, Forbes V, Gaya DR, Johnston BT, McKiernan PJ, Murray CD, Sebastian S, Smith M, Whitley L, Williams L, Russell RK, McCartney SA, Lindsay JO. UK guideline on transition of adolescent and young persons with chronic digestive diseases from paediatric to adult care. Gut. 2017 Jun;66(6):988-1000. doi: 10.1136/gutjnl-2016-313000. Epub 2017 Feb 21. PMID 28228488
- [Background] van Rheenen PF, Aloi M, Biron IA, Carlsen K, Cooney R, Cucchiara S, Cullen G, Escher JC, Kierkus J, Lindsay JO, Roma E, Russell RK, Sieczkowska-Golub J, Harbord M. European Crohn's and Colitis Organisation Topical Review on Transitional Care in Inflammatory Bowel Disease. J Crohns Colitis. 2017 Sep 1;11(9):1032-1038. doi: 10.1093/ecco-jcc/jjx010. PMID 28158494
- [Background] Suris JC, Akre C. Key elements for, and indicators of, a successful transition: an international Delphi study. J Adolesc Health. 2015 Jun;56(6):612-8. doi: 10.1016/j.jadohealth.2015.02.007. PMID 26003575
- [Background] Fair C, Cuttance J, Sharma N, Maslow G, Wiener L, Betz C, Porter J, McLaughlin S, Gilleland-Marchak J, Renwick A, Naranjo D, Jan S, Javalkar K, Ferris M; International and Interdisciplinary Health Care Transition Research Consortium. International and Interdisciplinary Identification of Health Care Transition Outcomes. JAMA Pediatr. 2016 Mar;170(3):205-11. doi: 10.1001/jamapediatrics.2015.3168. PMID 26619178
- [Background] van den Brink G, van Gaalen MAC, de Ridder L, van der Woude CJ, Escher JC. Health Care Transition Outcomes in Inflammatory Bowel Disease: A Multinational Delphi Study. J Crohns Colitis. 2019 Sep 19;13(9):1163-1172. doi: 10.1093/ecco-jcc/jjz044. PMID 30766997
- [Background] Eros A, Soos A, Hegyi P, Szakacs Z, Eross B, Parniczky A, Mezosi E, Rumbus Z, Sarlos P. Spotlight on Transition in Patients With Inflammatory Bowel Disease: A Systematic Review. Inflamm Bowel Dis. 2020 Feb 11;26(3):331-346. doi: 10.1093/ibd/izz173. PMID 31504524
- [Derived] Eros A, Dohos D, Veres G, Tarnok A, Vincze A, Teszas A, Zadori N, Gede N, Hegyi P, Sarlos P. Effect of joint transition visits on quality of life in adolescents with inflammatory bowel diseases: a protocol for a prospective, randomised, multicentre, controlled trial (TRANS-IBD). BMJ Open. 2020 Oct 6;10(10):e038410. doi: 10.1136/bmjopen-2020-038410. PMID 33028560